CLINICAL TRIAL: NCT04661657
Title: COvid-19 LongitUdinal Multiethnic BioImaging Assessment of CARDiovascular Sequelae (COLUMBIA CARDS) Registry
Brief Title: COvid-19 LongitUdinal Multiethnic BioImaging Assessment of CARDiovascular Sequelae Registry
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: AAAT0787
Record Dates: First submitted 2020-12-08; First posted 2020-12-10 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Covid19; Cardiac Disease; Cardiac Arrhythmia; Myocarditis; Left Ventricular Dysfunction
MeSH Terms: conditions — COVID-19; Heart Diseases; Arrhythmias, Cardiac; Myocarditis; Ventricular Dysfunction, Left | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19: Non-prisoner and non-pregnant subjects, without prior cardiac disease, who have tested positive or have been hospitalized due to COVID-19 infection. Subjects will be undergo a physical exam, blood draw to asses serological biomarkers. Subjects will also undergo an transthoracic echocardiogram (TTE) and a clariscan-enhanced cardiovascular magnetic resonance imaging (CMR) using a gadolinium based contrast agent (GBCA).
  Interventions: Other: Transthoracic echocardiogram (TTE); Other: Cardiovascular Magnetic Resonance (CMR) Imaging
- Control: Non-prisoner and non-pregnant subjects, without prior cardiac disease, who have never tested positive and/or has never been hospitalized due to COVID-19 infection. Subjects will be undergo a physical exam, blood draw to asses serological biomarkers. Subjects will also undergo an transthoracic echocardiogram (TTE) and a clariscan-enhanced cardiovascular magnetic resonance imaging (CMR) using a gadolinium based contrast agent (GBCA).
  Interventions: Other: Transthoracic echocardiogram (TTE); Other: Cardiovascular Magnetic Resonance (CMR) Imaging

INTERVENTIONS:
Other: Transthoracic echocardiogram (TTE) — Subjects will undergo TTE imaging.
Other: Cardiovascular Magnetic Resonance (CMR) Imaging — Subjects will undergo CMR Imaging using a gadolinium based contrast agent (GBCA).

SUMMARY:
COLUMBIA CARDS is a pilot study to understand how COVID-19 affects the heart. It is known that COVID-19 can affect the heart in different ways. COLUMBIA CARDS is studying why some COVID-19 survivors develop clinical conditions such as heart inflammation, fluid buildup, blood clots, and other cardiac problems during or after their COVID-19 illness, and why other ones do not. In this study, we will use cardiovascular magnetic resonance (CMR) and transthoracic echocardiography (TTE) to better understand the impact of COVID-19 on the heart.

DETAILED DESCRIPTION:
This is a pilot study aiming to collect preliminary data on cardiac imaging (CMR and TTE) in outpatients who recovered from COVID-19.

CMR offers the unique ability to comprehensively characterize myocardial tissue and assess the heart's structure and function, through a variety of complementary imaging techniques using different pulse sequences. The investigators propose to provide a multi-sequence CMR evaluation of a spectrum of convalescent COVID-19 patients, compare COVID-19 survivors to controls, and study the relationships between myocardial characteristics by CMR and echocardiography and health outcomes, and how these are modulated through patient characteristics, and clinical characteristics of COVID-19 illness. Broadly, this myocardial characterization will not just provide diagnosis but serve as a potentially powerful tool for risk stratification, therapeutic decision making, and monitoring response to therapies in COVID-19 survivors.

Transthoracic echocardiography (TTE) is the most widely used imaging technique for the assessment of cardiac morphology and function. While its capability for myocardial tissue characterization is inferior to that of CMR, TTE provides several advantages that make it an ideal complement to CMR for the assessment of cardiac involvement in COVID-19 patients. TTE offers a rapid noninvasive evaluation of myocardial and valvular function, in addition to the assessment of other cardiac abnormalities of interest (such as presence and amount of pericardial effusion) and important hemodynamic variables (noninvasive estimation of pulmonary pressures is an example). TTE is easily performed and reproducible, and does not involve the use of radiations or contrast agents, which allows the performance of repeat evaluations to assess serial changes over time in the cardiac parameters of interest.

ELIGIBILITY:
Inclusion Criteria:

* Convalescent COVID-19 patient
* If COVID-19 patient, at least 4 weeks after beginning of symptoms, and at least 2 weeks after hospital discharge if had been hospitalized.
* Control patients who have had a negative COVID-19 screening without prior positive tests.
* Willingness to undergo Clariscan-enhanced CMR scan.
* Ability to hold breath for 15 seconds.
* Willingness to give informed consent.
* Greater than or equal to 18 years of Age.

Exclusion Criteria:

* Subjects who are Pregnant or nursing
* Severe valvular heart disease
* History of congestive heart failure preceding COVID-19
* History of obstructive coronary artery disease with known stenosis >70% or fractional flow reserve < 0.8
* Contraindication to MRI
* Known allergy to gadoterate
* Estimated glomerular filtration rate <30 ml/min/1.73m2
* History of receiving more than 2 doses of a gadolinium-based contrast agent
* Subject is of prisoner status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age or older, without cardiac disease who have tested positive for COVID-19 or healthy control subjects who have not had COVID-19. Willing to undergo Cardiac MRI and Transthoracic echocardiogram. No known sensitivity to Gadolinium based contrast agent.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2022-01-22 (Actual)

PRIMARY OUTCOMES:
Percentage of myocardium demonstrating late gadolinium enhancement | Up to 2 hours
  Percentage of myocardium demonstrating late gadolinium enhancement by cardiac magnetic resonance (CMR) imaging, determined using Circle cvi42 software.
Extracellular Volume (ECV) Fraction | Up to 2 hours
  Extracellular volume fraction measured by CMR imaging. ECV determined using Circle cvi42 software and using formula ECV = (1-hematocrit) × (Δ(1/T1myocardium)/Δ(1/T1blood)).
Left Ventricular Ejection Fraction | Up to 2 hours
  Left ventricular ejection fraction (percent ejection fraction) by CMR imaging and determined using Circle cvi42 software.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Einstein, MD, PhD, Principal Investigator — Columbia Univeristy
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided